CLINICAL TRIAL: NCT02965404
Title: A Blind, Randomized and Controlled Clinical Trial to Evaluate the Safety of Live Attenuated Varicella Vaccines for Healthy Adults, Adolescents and Children
Brief Title: A Safety Study of Live Attenuated Varicella Vaccines in Healthy Adults, Adolescents and Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sinovac (Dalian) Vaccine Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO-VZV-1001
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2016-11

CONDITIONS: Varicella
Keywords: live attenuated varicella vaccine; safety; adult; adolescent; child
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Experimental Group (Experimental): * Single intramuscular injection of the investigational vaccine (0.5 ml) on Day 0;
  * Intervention: investigational live attenuated varicella vaccine.
  Interventions: Biological: Investigational live attenuated varicella vaccine
- Positive Control Group (Active Comparator): * Single intramuscular injection of the control vaccine (0.5 ml) on Day 0;
  * Intervention: control live attenuated varicella vaccine.
  Interventions: Biological: control live attenuated varicella vaccine
- Negative Control Group (Sham Comparator): * Single intramuscular injection of the diluent of lyophilized vaccine (0.5 ml) on Day 0;
  * Intervention: diluent of lyophilized vaccine.
  Interventions: Biological: diluent of lyophilized vaccine

INTERVENTIONS:
Biological: Investigational live attenuated varicella vaccine — The investigational vaccine was manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd.
  Arms: Experimental Group
Biological: control live attenuated varicella vaccine — The control vaccine was manufactured by Shanghai Institute of Biological Products Co., Ltd. (SIBP)
  Arms: Positive Control Group
Biological: diluent of lyophilized vaccine — The diluent of lyophilized vaccine was manufactured by Sinovac (Dalian) Vaccine Technology
  Arms: Negative Control Group

SUMMARY:
The purpose of this study is to evaluate the safety of a live attenuated varicella vaccine in healthy adults, adolescents, and children.

DETAILED DESCRIPTION:
This study is a randomized, blind, single-center, controlled phase I clinical trial. The purpose of this study is to evaluate the safety of a live attenuated varicella vaccine manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd. The positive control is a commercialized live attenuated varicella vaccine manufactured by Shanghai Institute of Biological Products Co., Ltd. (SIBP), and the negative control is diluent of lyophilized vaccine manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd. All participants are healthy, and will be randomly assigned into experimental group, positive control group, or negative control group in the ratio 1:1:1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer between 1 - 49 years old;
* Proven legal identity;
* Guardian(s) of the volunteer and/or volunteers themselves should be capable of understanding the written consent form, and such form should be signed before the infant being included into this study;

Exclusion Criteria:

* Prior vaccination with varicella vaccine or with history of varicella zoster virus (VZV) infection;
* Axillaty temperature > 37.0 °C;
* Breast feeding, pregnant, or expected to conceive during the period of this trial;
* History of allergy to any vaccine or vaccine ingredient, or serious adverse reaction(s) to vaccination, such as urticaria, difficulty in breathing, angioneurotic edema, abdominal pain, etc;
* History of epilepsy, seizures or convulsions, or a family history of mental illness;
* Autoimmune disease or immunodeficiency;
* Severe malnutrition, congenital malformation, developmental disorders, or serious chronic diseases;
* Acute disease or acute stage of chronic disease within 7 days prior to study entry;
* Receipt of any of the following products:

  1. Any subunit vaccine or inactivated vaccine within 7 days prior to study entry;
  2. Any live attenuated vaccine within 1 month prior to study entry;
  3. Any blood product, immunosuppressant, hormone, or other investigational medicine(s) within 30 days prior to study entry;
* Any significant abnormity of heart, lung, skin, or pharynx;
* Any of the pre-immune test results of the following indexes of laboratory tests showed clinically significant abnormity:

  1. Blood routine examinations: hemoglobin (Hb), white blood cells (WBC) count;
  2. Blood biochemistry detections: alanine transferase (ALT), total bilirubin, blood urea nitrogen (BUN), creatinine;
  3. Urine routine tests: urine protein, urine glucose, urine erythrocyte
* Any other factor that suggesting the volunteer is unsuitable for this study based on the opinions of investigators;

Ages: 1 Year to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 270 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The incidences of adverse events (AEs) of each group | 30 days
  AEs occurred within 30 days after injection will be collected.

SECONDARY OUTCOMES:
The incidences of abnormal results of lab tests | 30 days
  Cases of abnormal results of laboratory tests will be collected.
The incidences of serious adverse events (SAEs) of each group | 30 days
  SAEs occurred within 30 days after injection will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Shengli Xia, Principal Investigator — Henan Provincial Center for Disease Control and Prevention
Locations (1):
- Xiangcheng County Center for Disease Control and Prevention, Xuchang, Henan, China

IPD SHARING:
Plan to Share IPD: No